CLINICAL TRIAL: NCT00426179
Title: An Exploratory Study of the Effects of Imatinib on Allergic Inflammation Following Out of Allergy Season Repeated Nasal Allergen Challenge in Subjects With Seasonal Allergic Rhinitis Sensitive to Timothy Grass Pollen - an Exploratory Study of c-Kit Inhibition in Allergic Respiratory Diseases
Brief Title: Effects of Imatinib in Subjects With Seasonal Allergic Rhinitis and Who Are Sensitive to Timothy Grass Pollen
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSTI571E2204
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-11

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Imatinib, allergic inflammation, out of allergy season, repeated nasal allergen, seasonal allergic rhinitis, sensitive, Timothy grass pollen, c-kit inhibition
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib

SUMMARY:
This study will assess the effects of Imatinib on allergic inflammation following repeated nasal allergen challenge in subjects with seasonal allergic rhinitis sensitive to Timothy grass pollen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male non-smoking subjects aged 18-55 years, with a history of seasonal allergic rhinitis consistent with Timothy grass pollen allergy. They must show: a positive skin prick test to Timothy grass pollen (wheal difference Timothy grass pollen - negative control ≥ 3 mm) at or within the 12 months preceding the screening visit and demonstrate symptomatic worsening (TNSS ≥4) within one hour after nasal allergen challenge
* Be otherwise healthy with no health problems that may jeopardize the subjects participating in the study, absence of history of other significant allergies.
* Subjects and their partners must agree to use effective contraceptive measures from screening until the end of study visit.

Exclusion Criteria:

* Respiratory disease other than a history of mild stable asthma not requiring treatment and associated with normal lung function.
* Structural nasal abnormalities or nasal polyps on examination, a history of frequent nose bleeding, recent nasal surgery or recent (within 8 weeks prior to baseline visit) or recent (four weeks) or ongoing upper or lower respiratory tract infection.
* Use of any medication that would affect the response to the allergen challenge (e.g. corticosteroids, decongestants, anti-histamines, medications with anti-inflammatory effects) or any other nasally applied medication within 14 days prior to allergen challenge (30 days for systemic anti-inflammatory therapy including oral corticosteroids), or known to influence Imatinib bioavailability or clearance
* History or laboratory evidence of acute or chronic renal insufficiency or abnormal liver function.
* Subjects may voluntarily withdraw from or be withdrawn from the study at the discretion of the investigator or the sponsor at any time. Subjects may be withdrawn from the study prematurely for one of the following reasons:
* Subject withdrew consent
* Upper respiratory tract infection
* Presence of allergic rhinitis symptoms in the screening period or prior to pre-wash on Day 1
* A past medical history of inherited heart disease, valve defect, cardiomyopathy, rheumatic fever, arrhythmias, cardiac interventions or clinically significant ECG abnormalities.
* Adverse events and non-tolerable symptoms resulting from allergen challenge
* Administration of a concomitant medication (other than those randomized to receive Fluticasone propionate) that would impact on the study results (e.g. corticosteroids), including any subjects requiring asthma therapy (inhaled or systemic).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-12; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Effect of Imatinib on the reduction of mast cell degranulation (measured by β-tryptase and PGD2) in response to allergen challenge

SECONDARY OUTCOMES:
Additional markers of inflammation following nasal allergen challenge (NAC):
Enumeration of eosinophils in nasal lavage following NAC
Total nasal symptom score (TNSS) following NAC
Soluble mediators collected from adsorption onto nasal filter papers following NAC, with a focus on Th2-associated cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis Investigative site, Horsham, United Kingdom